CLINICAL TRIAL: NCT01773590
Title: Mechanisms of Interplay Between Allergy and Viruses in Asthma: A Human Model of Rhinovirus Induced Acute Asthma Exacerbations
Brief Title: Mechanisms of Interplay Between Allergy and Viruses in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12/LO/1278; 12/LO/1278 (Other: London Bridge Research Ethics Commitee)
Record Dates: First submitted 2012-11-30; First posted 2013-01-23 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Rhinovirus Infection in Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asthmatics (Other): Rhinovirus Infection
  Interventions: Other: Rhinovirus Infection
- Healthy Volunteers (Other): Rhinovirus Infection
  Interventions: Other: Rhinovirus Infection

INTERVENTIONS:
Other: Rhinovirus Infection

SUMMARY:
The aim of this study is to investigate the mechanisms of interplay between allergy (IgE and Th2 mediated inflammation) and virus infection in the development of asthma, as well as the risk and severity of acute exacerbations of asthma. Understanding these mechanisms should identify new approaches for novel therapies for the prevention of asthma development and for prevention/treatment of asthma exacerbations. Such treatment has potential to have a major impact on patient quality of life and to result in enormous reductions in health care costs.

A human model will be used to identify dysregulated genes/proteins and determine relationships with disease outcomes. This study will compare lower airway responses between asthmatic and healthy control subjects undergoing rhinovirus (RV) experimental infection (subjects will be infected with rhinovirus as part of the study). This will have the dual advantage of investigating mechanisms in the most natural model possible, as well as developing a better model for testing novel therapeutic approaches. The investigators will analyse the samples from both subject groups, to determine their relevance to the human disease. Any genes/proteins shown to be dysregulated and related to disease outcomes in the human model will be very strong candidates for immediate translation into human intervention studies.

Up to 12 asthmatic and/or healthy subjects will be recruited for a preliminary pilot study. These subjects will be ineligible to enter the main study due to the presence of neutralizing antibody to RV16 (~50% of subjects otherwise suitable for the study). These subjects will meet all other inclusion/exclusion criteria for the main study. The 12 participants will undergo tests including a single bronchoscopy, nasal sampling and blood tests allowing for optimisation of all sample processing techniques. They will not be infected with RV-16.

In the main study the investigators will aim to study up to 15 healthy volunteers and 15 volunteers with moderate asthma (all on inhaled steroid treatment). Subjects will undergo a single baseline bronchoscopy 2 weeks prior to inoculation with the RV16 virus. Following infection with the virus participants will be required to attend for regular sample collection including 2 further bronchoscopies post-infection. Patients will be followed until convalescence 6 weeks post infection.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for Asthmatic subjects:

* Age 18-55 years
* Doctor diagnosis of Asthma
* Histamine PC20 < 8 µg/ml (or <12 µg/ml and bronchodilator response ≥ 12%) and worsening asthma symptoms with infection since last change in asthma therapy
* Atopic on skin testing
* Treatment comprising ICS or combination inhaler (LABA+ICS)

  *subjects on inhaled corticosteroids must be on a daily dose of 400mcg fluticasone or equivalent.
* An Asthma Control Questionnaire (ACQ) score of > 0.75.

Inclusion criteria for healthy controls:

* Age 18-55 years
* No history or clinical diagnosis of asthma
* No history of allergic rhinitis or eczema
* Negative responses on skin prick testing
* PC20 > 8 µg/ml and bronchodilator response <12%
* Absence of current or previous history of significant respiratory disease
* Absence of significant systemic disease

Exclusion Criteria:

Exclusion criteria for Asthmatic subjects:

* Smoking history over past 6 months
* Negative skin prick tests
* Current symptoms of allergic rhinitis
* Current or previous history of significant respiratory disease (other than asthma)
* Any clinically relevant abnormality on screening or detected significant systemic disease
* Pregnant or breastfeeding women
* Contact with infants or elderly at home or at work
* Asthma exacerbation or viral illness within the previous 6 weeks
* Treatment with oral steroids now or in the previous 3 months
* Current use of nasal spray, anti-histamine, anti-leukotrienes
* Antibodies to rhinovirus 16 in a titre >1:2

Exclusion criteria for healthy controls:

* Any clinically relevant abnormality on screening or detected significant systemic disease
* A current or previous diagnosis of asthma
* Any positive skin prick test
* Current symptoms of allergic rhinitis
* History of eczema or allergic rhinitis
* Pregnant or nursing women
* Common cold within the previous 8 weeks
* Treatment with oral or inhaled steroids now or in the previous 3 months; current use of long-acting β-agonists, nasal spray, anti-histamine, leukotrienes or tiotropium.
* Shortness of breath score at screening over 1 or total lower respiratory tract score over 7
* Antibodies to rhinovirus 16 in a titre >1:2

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2013-02; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Host response to RV challenge | Prior to and 0-42 days post challenge
  The host response to RV challenge will be assessed daily for 8 days using methods including symptom diaries, lung function, detection of mediators in nasal and bronchial lining fluid, characterisation of different cell types in bronchoalveolar lavage as determined by flow cytometry. This will be compared with findings at baseline, day 11, 15 and up to 42 days post challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Johnston, Principal Investigator — National Heart and Lung Institute
Locations (1):
- National Heart and Lung Institute, London, London, United Kingdom